CLINICAL TRIAL: NCT00333944
Title: Effectiveness of High Dose Pralidoxime in the Treatment of Organophosphorus Pesticide Poisoning - a Randomised Controlled Trial
Brief Title: Study to Know the Efficacy of Higher Doses of Pralidoxime in Patients of Organophpsphorus Poisoning.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giriraj Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GRH/IERC/2000/12
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2006-06-06 (Estimated); Status verified 2000-05

CONDITIONS: Acute Organophosphorus Pesticide Poisoning
Keywords: Organophosphorus poisoning; Atropine; Pralidoxime; Intermediate syndrome.
MeSH Terms: conditions — Organophosphate Poisoning | interventions — atropine, pralidoxime iodide, trichlorofon drug combination

INTERVENTIONS:
Drug: Pralidoxime(drug)

SUMMARY:
The purpose of this study is to determine whether high doses of pralidoxime(PAM) are effective as compare to lower doses of PAM in the management of moderately sever organophosphorus poisoning patients.

DETAILED DESCRIPTION:
Standard treatment of organophosphorus pesticide poisoning involves administration of intravenous atropine and oximes to counter acetylcholinesterase inhibition.1 Treatment with atropine is well established, but the efficacy and dosage schedule of oximes are controversial.2-5 A dose of 1g every four to six hours has been the standard regimen in Asian district hospitals but many clinicians remain unconvinced by its effectiveness.3 Randomised controlled trials (RCT) performed in Vellore during the nineties compared a 12g infusion over 3-4 days with a 1g bolus dose and then with placebo.6,7 The authors reported no benefit from pralidoxime and an increased mortality in those receiving the infusion, and have stated that pralidoxime should not be given to organophosphorus poisoned patients.2

Others consider that the dosage regimen was not ideal, with therapeutic concentrations being obtained rarely during the treatment.3,4 Furthermore, many patients presented late and had taken dimethyl pesticides - a class that does not respond well to oximes after several hours - biasing the study against finding benefit.

The proposed minimum effective plasma levels for pralidoxime of 4 mg/L were based on in vitro and animal experiments by Sundwall.8 Recent evidence, however, suggests that higher blood concentrations of pralidoxime are needed to antagonise the toxic effects of many pesticides and that a bolus loading infusion followed by a maintenance infusion would be the best regimen.9 The WHO have proposed that patients receive around 30mg/kg pralidoxime salt as a loading dose followed by an infusion of at least 8mg/kg/hr (roughly equivalent to 1-2 g bolus followed by 0·5 g/h in a 50kg south Asian patient).9,10 However, no trials have yet been performed to determine whether such a regimen reduces morbidity and mortality in severely poisoned patients.3 Since organophosphorus pesticides kill hundreds of thousands of people in rural Asia every year, it is essential to determine whether it benefits or harms such poisoned patients.

Our hospital has typically used a regimen of 1g q4h in organophosphorus poisoned patients but we were unconvinced about the effectiveness of this expensive drug since many patients required ventilation for >10 days. We informally treated several patients with the WHO-recommended regimen but saw little benefit. Since pralidoxime has a high therapeutic index, we then decided to conduct a RCT with still higher doses, i.e. to compare a 1 g infusion every hour (q1h, 24 g/day) with 1g every four hours (q4h, 6 g/day), after a 2 g loading dose, to assess the effectiveness of high dose pralidoxime in organophosphorus poisoned patients.

ELIGIBILITY:
Inclusion Criteria:

-patients with a history of poisoning by an organophosphorus pesticide and clinical features of poisoning.

Exclusion Criteria:

patients who

* were under 12 years
* had chronic disease
* had malignancy
* were pregnant,
* presented more than 24 hrs post-ingestion,
* who could not be resuscitated successfully in the emergency room of our ospital

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2000-05; Study Completion 2003-06

PRIMARY OUTCOMES:
Median atropine dose required in first 24 hours
proportion of patients who required intubation or developed intermediate syndrome
number of days ventilated and required ICU care

SECONDARY OUTCOMES:
pneumonia (aspiration or ventilator-associated)
mean systolic and diastolic blood pressure (BP) in first 24 hours
case fatality

CONTACTS AND LOCATIONS:
Overall Officials: Kirti S Pawar, MBBS,DA, Principal Investigator
Locations (1):
- Giriraj Hospital and Intensive Care Unit., Baramati. Pune District., Maharashtra, India

REFERENCES:
- [Derived] Pawar KS, Bhoite RR, Pillay CP, Chavan SC, Malshikare DS, Garad SG. Continuous pralidoxime infusion versus repeated bolus injection to treat organophosphorus pesticide poisoning: a randomised controlled trial. Lancet. 2006 Dec 16;368(9553):2136-41. doi: 10.1016/S0140-6736(06)69862-0. PMID 17174705